CLINICAL TRIAL: NCT05761821
Title: Relationship Between Key Factors of Leadless Pacemaker Implantation With Implantation Site, Intraoperative Complications and Prognosis
Brief Title: Key Factors of Leadless Pacemaker Implantation With Implantation Site, Complications and Prognosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yangxin Chen, Chief physician, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSKY-2023-056-01
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-02

CONDITIONS: Complication of Surgical Procedure; Pacemaker Complication; Pacemaker Syndrome
Keywords: leadless pacemaker; complication; Prognosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Leadless pacemaker — All enrolled patients were implanted with leadless pacemaker.

SUMMARY:
To investigate the relationship between key variables in leadless pacemaker implantation with implantation site, intraoperative complications and prognosis.

DETAILED DESCRIPTION:
In this study, we aim to include patients implated with leadless pacemakers, collect key variables and other clinical data during implantation of leadless pacemakers, and observe the final implantation site, intraoperative complications and prognosis information of patients. This study aims to clarify the relationship between key variables in leadless pacemaker implantation with implantation site, intraoperative complications and prognosis, and provide data support for the standardization of leadless pacemaker implantation process in China.

ELIGIBILITY:
Inclusion Criteria:

* Patient received implantation of leadless pacemaker
* Patient agreed to join into this study and signed informed consent

Exclusion Criteria:

* Age < 18 years
* Ventricular septal defect
* History of mechanical tricuspid valve replacement
* History of inferior vena cava filter placement
* Pregnant or plan to be pregnant within 2 years
* Life expectancy < 1 year
* Patient was included in other studies that could introduce bias into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients received implantation of leadless pacemaker
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Serious adverse events | Day 0 (Time of implantation)-Day 7
  including dislodgement (including detachment), cardiac perforation, pericardial effusion, and serious infection

SECONDARY OUTCOMES:
Device-related complications | Day 0 (Time of implantation)-Day 7
  Femoral venipuncture site hematoma, hemorrhage, pseudoaneurysm, arteriovenous fistula, tricuspid valve injury
Device-related complications | Day 0 (Time of implantation)-Year 2
  Femoral venipuncture site hematoma, hemorrhage, pseudoaneurysm, arteriovenous
Serious adverse events | Day 0 (Time of implantation)-Year 2
  including dislodgement (including detachment), cardiac perforation, pericardial effusion, and serious infection
Re-intervention of devices | Day 0 (Time of implantation)-Year 2
  extraction, re-implantation, or implantation of traditional transvenous pacemaker

CONTACTS AND LOCATIONS:
Overall Officials: Yangxin Chen, PhD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided